CLINICAL TRIAL: NCT01339442
Title: A Phase 1 Trial of BKM 120, a Novel Oral Selective Phosphatidylinositol-3-kinase (PI3K) Inhibitor, in Combination With Fulvestrant in Postmenopausal Women With Estrogen Receptor Positive Metastatic Breast Cancer
Brief Title: BKM120 and Fulvestrant for Treating Postmenopausal Patients With Estrogen Receptor-Positive Stage IV Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201105445; NCI-2011-00583 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-04-13; First posted 2011-04-20 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Estrogen Receptor-positive Breast Cancer; Recurrent Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — NVP-BKM120; Fulvestrant; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Level 1 - Phase 1A (Experimental): BKM120 80 mg PO daily.
  Fulvestrant 500 mg IM on Days 1 & Day 15 during Cycle 1 then on Day 1 of each subsequent cycle.
  Interventions: Drug: BKM120; Drug: Fulvestrant; Procedure: biopsy
- Dose Level 2 - Phase IA (Experimental): BKM120 100 mg PO daily.
  Fulvestrant 500 mg IM on Days 1 & Day 15 during Cycle 1 then on Day 1 of each subsequent cycle.
  Interventions: Drug: BKM120; Drug: Fulvestrant; Procedure: biopsy
- Phase IB (Experimental): BKM120 (dose to be determined in Phase IA)PO 5 days on/ 2 days off per week.
  Fulvestrant 500 mg IM on Days 1 & Day 15 during Cycle 1 then on Day 1 of each subsequent cycle.
  Interventions: Drug: BKM120; Drug: Fulvestrant; Procedure: biopsy
- Cohort C (Experimental): BKM120 (dose determined in Phase IA) PO daily.
  Fulvestrant 500 mg IM on Day 1 and Day 15 during Cycle 1 then monthly on Day 1 of subsequent cycles.
  Interventions: Drug: BKM120; Drug: Fulvestrant; Procedure: biopsy

INTERVENTIONS:
Drug: BKM120
  Other Names: PI3K_Inhibitor_BKM120
Drug: Fulvestrant
  Other Names: Faslodex; ICI 182,780
Procedure: biopsy — Correlative studies
  Other Names: biopsies

SUMMARY:
This phase I trial will determine the Maximum Tolerated Dose (MTD) of BKM120 when given together with fulvestrant in treating postmenopausal patients with estrogen receptor-positive (ER+) stage IV breast cancer. The toxicity profile of this combination therapy will also be described. Inhibition of PI3K by BKM120 may enhance programmed cell death (apoptosis) in estrogen receptor positive (ER+) breast cancer cells. Giving fulvestrant together with BKM 120 may enhance this apoptotic effect, providing a novel therapeutic strategy for patients with metastatic ER+ breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of BKM120 (PI3K inhibitor BKM120) in combination with fulvestrant.

II. To evaluate the toxicity profile of BKM120 in combination with fulvestrant.

SECONDARY OBJECTIVES:

I. To evaluate the toxicity profile of BKM120 in combination with fulvestrant when administered for at least 3 months.

II. To determine the steady state blood concentrations of BKM120 when combined with fulvestrant.

III. To evaluate the anti-tumor effect (partial response [PR], complete response [CR], stable disease [SD], and progressive disease [PD]) of BKM120 in combination with fulvestrant in patients with ER+ metastatic breast cancer.

TERTIARY OBJECTIVES:

I. To examine baseline tumor specimens for phosphatidylinositol 3-kinase (PI3K) pathway abnormalities, and to correlate with treatment response.

II. To examine the PIK3 catalytic alpha polypeptide (PIK3CA) mutation status in circulating deoxyribonucleic acid (DNA) at baseline and following study therapy and to correlate with tumor tissue PIK3CA status and treatment response.

III. To determine effects of study therapy on fasting C-peptide and glucose. IV. To evaluate target inhibition by BKM120 on serial tumor biopsies collected before and following study therapy.

V. To evaluate the effect of BKM120 in combination with fulvestrant on tumor cell proliferation and apoptosis.

VI. To obtain preliminary pilot data to evaluate the effect of BKM120 on tumor cell proliferation, as measured by FLT-PET/CT (Phase IB)

OUTLINE: This is a dose-escalation study of PI3K inhibitor BKM120. Patients receive PI3K inhibitor BKM120 orally (PO) once daily (QD) on days 1-28 (if enrolled in Phase IA or Cohort C) or on a 5 days on/2 days off schedule (if enrolled in Phase IB). All patients will receive fulvestrant intramuscularly (IM) on days 1 and 15 of Cycle 1 and day 1 of all subsequent cycles. Cycles repeat ever 28 days in the absence of disease progression or unacceptable toxicity.

Two OPTIONAL FLT-PET/CT scans: the first one done at baseline before the start of BKM120 and the second one done between Day 16 and Day18 after BKM120 is started. After completion of study treatment, patients are followed up for 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be ≥ 18 years of age
* Patient must be a postmenopausal woman, defined by one of the following criteria:

  * Women ≥ 60 years
  * Women aged 45-59 years with spontaneous cessation of menses ≥ 12 months prior to registration
  * Women aged 45-59 years with cessation of menses of duration < 12 months or secondary to hysterectomy AND an follicle-stimulating hormone (FSH) level in the postmenopausal range according to institutional standards (or > 34.4 IU/L if institutional range is not available) prior to registration
  * Women aged 45-59 years on hormonal replacement therapy who have discontinued hormonal therapy AND an FSH level in the postmenopausal range according to institutional standards (or > 34.4 IU/L if institutional range is not available) prior to registration
  * Status post bilateral surgical oophorectomy
* Patient must have a negative serum pregnancy test within 48 hours before starting study treatment (if a woman of childbearing potential)
* Patient must have an Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Patient must have histologically or cytologically confirmed invasive breast cancer that is stage IV or metastatic (histologic/cytologic confirmation of recurrence preferred, but not required)
* Patient must have a representative tumor tissue specimen available; archival tissue is allowed
* Either the primary or the metastatic tumor must be positive for estrogen receptor (>= 1% tumor cell staining by immunohistochemistry or an Allred Score of >= 3 by immunohistochemistry)
* Patient must have at least one site of measurable disease as per Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 criteria
* Patient must have had no more than 3 lines of systemic therapy (including endocrine therapy) for metastatic disease to be eligible for phase IB and the last 10 patients of Cohort C; there is no limitation on the numbers of prior systemic therapies for phase IA and the first 2 patients of Cohort C
* Patients who are currently taking fulvestrant without disease progression are eligible
* Patient must have a life expectancy of >= 12 weeks
* Patient must have adequate oran function as defined as:

  * Absolute neutrophil count (ANC) >= 1500/uL
  * Platelet count >= 100,000/uL
  * Hemoglobin >= 9 g/dL
  * Serum creatinine =< 1.5 x upper limit of normal (ULN)
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) within normal range (or =< 3.0 x ULN if liver metastases are present)
  * Serum bilirubin =< ULN (or =< 1.5 x ULN if liver metastases are present; or total bilirubin =< 3.0 x ULN with direct bilirubin within normal range in patients with well documented Gilbert Syndrome)
  * Serum amylase =< ULN
  * Serum lipase =< ULN
  * Magnesium >= the lower limit of normal
  * Potassium within normal limits for the institution
* Patient must have international normalized ratio (INR) =< 2
* Patient must have fasting plasma glucose =< 120 mg/dL (6.7 mmol/L)
* Patient must have total calcium (corrected for serum albumin) within normal limits (bisphosphonate use for malignant hypercalcemia control is not allowed)
* Patient must be able and willing to sign the consent form

Exclusion Criteria:

* Patient must not have received prior treatment with a P13K inhibitor
* Patient must not have a known hypersensitivity to BKM120 or to its excipients
* Patient must not have untreated brain metastases; however, patients with metastatic central nervous system (CNS) tumors may participate in this trial if the patient is:

  * 4 weeks from therapy completion (including radiation and/or surgery)
  * Clinically stable at the time of study entry
  * Not receiving corticosteroid therapy
* Patient must not have acute or chronic liver disease, renal disease, or pancreatitis
* Patient must not have any of the following mood disorders as judged by the Investigator or a Psychiatrist

  * Medically documented history of or active major depressive episode, bipolar disorder (I or II), obsessive-compulsive disorder, schizophrenia, a history of suicidal attempt or ideation, or homicidal ideation (immediate risk of doing harm to others)
  * Greater than or equal to Common Terminology Criteria for Adverse Events (CTCAE) grade 3 anxiety
* Patient must not meet the cut-off score of >= 10 in the Patient Health Questionnaire (PHQ-9) or a cut-off of >= 15 in the Generalized Anxiety Disorder (GAD)-7 mood scale, respectively, or select a positive response of 1, 2, or 3 to question number 9 regarding potential for suicidal thoughts in the PHQ-9 (independent of the total score of the PHQ-9)
* Patient must not have >= grade 2 diarrhea
* Patient must not have active cardiac disease including any of the following:

  * Left ventricular ejection fraction (LVEF) < 50% as determined by Multiple Grated acquisition (MUGA) scan or echocardiogram (ECHO)
  * QTc > 480 msec on screening electrocardiogram (ECG) (using the QTcF formula)
  * Angina pectoris that requires the use of anti-anginal medication
  * Ventricular arrhythmias except for benign premature ventricular contractions
  * Supraventricular and nodal arrhythmias requiring a pacemaker or not controlled with medication
  * Conduction abnormality requiring a pacemaker
  * Valvular disease with document compromise in cardiac function
  * Symptomatic pericarditis
* Patient must not have a history of cardiac dysfunction including any of the following:

  * Myocardial infarction within the last 6 months, documented by persistent elevated cardiac enzymes or persistent regional wall abnormalities on assessment of LVEF function
  * History of documented congestive heart failure (New York Heart Association functional classification III-IV)
  * Documented cardiomyopathy
* Patient must not have poorly controlled diabetes mellitus or steroid-induced diabetes mellitus (defined by fasting glucose >120 mg/dL or hemoglobin [Hb] A1c > 7%)
* Patient must not have any other concurrent severe and/or uncontrolled concomitant medical conditions (e.g., active or uncontrolled infection) that could cause unacceptable safety risks or compromise compliance with the protocol
* Patient must not have significant symptomatic deterioration of lung function; if clinically indicated, pulmonary function tests including measures of predicted lung volumes; diffusion capacity of carbon monoxide (DLco), oxygen (O2) saturation at rest on room air should be considered to exclude pneumonitis or pulmonary infiltrates
* Patient must not have impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of BKM120 (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection); patients with unresolved diarrhea will be excluded as previously indicated
* Patient must not have been treated with any hematopoietic colony-stimulating growth factors (e.g., filgrastim [G-CSF], sargramostim [GM-CSF]) =< 2 weeks prior to starting study drug; erythropoietin or darbepoetin therapy, if initiated at least 2 weeks prior to enrollment, may be continued
* Patient must not have taken herbal medications and certain fruits within 7 days prior to starting study drug; herbal medications include, but are not limited to: St. Johns wort, Kava, ephedra (ma huang), gingko biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, and ginseng; fruits include the CYP3A inhibitors Seville oranges, grapefruit, pummelos, or exotic citrus fruits
* Patient must not be currently receiving treatment with medication with a known risk to prolong the QT interval or inducing Torsades de Pointes unless the treatment can either be discontinued or switched to a different medication prior to starting study drug; please refer to Table 5-2 for a list of prohibited QT prolonging drugs with risk of Torsades de Pointes
* Patient must not be receiving chronic treatment with steroids or another immunosuppressive agent; Note: topical applications (e.g. rash), inhaled sprays (e.g. obstructive airways diseases), eye drops or local injections (e.g. intra-articular) are allowed; patients with previously treated brain metastases who are on stable low dose corticosteroids treatment (e.g. dexamethasone 2 mg/day, prednisolone 10 mg/day) for at least 14 days before start of study treatment are eligible
* Patient must not be currently treated with drugs known to be moderate or strong inhibitors or inducers of isoenzyme cytochrome P450, family 3, subfamily A (CYP3A) unless the treatment can be discontinued or switched to a different medication prior to starting study drug (please note that co-treatment with weak inhibitors of CYP3A is allowed)
* Patient must not have received chemotherapy or targeted anticancer therapy =< 4 weeks (6 weeks for nitrosourea, antibodies or mitomycin-C) prior to starting study drug
* Patient with any residual toxicities may not be enrolled unless all toxicities recover to =< grade 1 before starting the trial
* Patient must not have received any continuous or intermittent small molecule therapeutics (excluding monoclonal antibodies) =< 5 effective half lives prior to starting study drug; patient must have recovered from side effects of such therapy
* Patient must not have received wide field radiotherapy =< 4 weeks or limited field radiation for palliation =< 2 weeks prior to starting study drug; patient must have recovered from side effects of such therapy
* Patient must not have undergone major surgery =< 2 weeks prior to starting study drug; patient must have recovered from side effects of such therapy
* Patient must not be currently taking therapeutic doses of warfarin sodium or any other Coumadin-derivative anticoagulant
* Patient must not have a known diagnosis of human immunodeficiency virus (HIV) infection
* Patient must not have a history of another malignancy within 3 years, except cured basal cell carcinoma of the skin or excised carcinoma in situ of the cervix

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2011-11-14 (Actual); Primary Completion 2016-12-21 (Actual); Study Completion 2016-12-28 (Actual)

PRIMARY OUTCOMES:
MTD of BKM120 in combination with fulvestrant | 28 days (completion of cycle 1)
  Highest dose level at which no more than 1 of 6 patients develops a dose-limiting toxicity
Number of participants with adverse events after treatment with BKM120 in combination with fulvestrant | 28 days after completion of treatment

SECONDARY OUTCOMES:
Anti-tumor effect (PR, CR, SD and PD) of BKM120 in combination with fulvestrant | End of treatment (approximately 3 months)
Steady state blood concentration of BKM120 | Baseline, Cycle 2 Day 1, Cycle 3 Day 1
Tumor PI3K pathway abnormalities in tissue from previous biopsy or collected at baseline | Baseline
Effects of study therapy on blood levels of fasting C-peptide | Baseline, Cycle 1 Day 1, Cycle 2 Day 1, Cycle 3 Day 1
Effects of study therapy on blood levels of glucose | Baseline, Cycle 1 Day 1, Cycle 1 Day 15, Cycle 2 Day 1, Cycle 2 Day 15, Cycle 3 Day 1, End of Treatment
Samples will be analyzed for markers of PI3K signaling (including pAKT, pS6, Cyclin D1, subcellular localization of FOXO3a, phosphoproteomics), tumor cell proliferation (Ki67) and apoptosis (cleaved caspase 3 or TUNEL staining). | Baseline
Examine the PIK3CA mutation status in circulating DNA at baseline thru last treatment | Baseline or Cycle 1 Day 1 and Day 1 of each subsequent cycle

OTHER OUTCOMES:
FLT-PET/CT effect of BKM120 on tumor cell proliferation | 18 days
  To obtain preliminary pilot data to evaluate the effect of BKM120 on tumor cell proliferation, as measured by FLT-PET/CT

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Ma, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu